CLINICAL TRIAL: NCT02917135
Title: European Angel® Catheter Post Market Registry
Brief Title: Angel® Catheter Post Market Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: BiO2 Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: QD-180
Record Dates: First submitted 2016-09-23; First posted 2016-09-28 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-10

CONDITIONS: Pulmonary Embolism; Medical Device Complication; Deep Vein Thrombosis; Catheter Thrombosis; Catheter-related Bloodstream Infection (CRBSI) Nos
MeSH Terms: conditions — Pulmonary Embolism; Venous Thrombosis; Pyloric Stenosis, Hypertrophic

STUDY DESIGN:
Observational Model: Case-Only
Patient Registry: Yes
Target Follow-Up Duration: 33 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Angel® Catheter: All consecutive, hospitalized patients in whom the Angel® Catheter is placed, or there has been an attempt to place, at selected Registry sites.
  Interventions: Device: Angel® Catheter

INTERVENTIONS:
Device: Angel® Catheter — The Angel® Catheter is a retrievable inferior vena cava (IVC) filter attached to a multi-lumen central venous access (CVC) catheter. The device is designed to be placed at the bedside in the inferior vena cava, via the femoral vein, for the prevention of pulmonary embolism (PE) and for access to the central venous system.
  The Angel® Catheter is intended for short-term (less than 30 days) vascular access via the femoral vein.

SUMMARY:
This is a post-market, observational, retrospective multi-center Registry designed to gather information on the performance of the Angel® Catheter in general clinical practice.

DETAILED DESCRIPTION:
The Registry population will include all consecutive patients in whom the Angel® Catheter is placed at participating sites. Information about the use of the catheter will be collected from placement through three days after device removal, or through death or discharge, whichever occurs first. Date of discharge/transfer from the Critical Care Unit will also be collected, completing the defined registry observation.

Information on up to 2,000 patients will be abstracted from a patient chart review. Sites will be asked to record data on all Angel® Catheter placements in their institution starting with their first Angel® Catheter placement after training by BiO2 Medical, Inc. personnel once all necessary institutional approvals are obtained confirming that Informed Consent is not required from the patient or LAR to collect, use, or publish patient data from this registry.

The registry population will include all consecutive patients in whom the Angel® Catheter is placed, or there has been an attempt to place, at selected Registry sites. The Instructions for Use (IFU) for the Angel® Catheter include the following indications:

* Pulmonary thromboembolism when anticoagulants are contraindicated; or
* Failure of anticoagulant therapy in thromboembolic diseases; or
* Emergency treatment following massive pulmonary embolism where anticipated benefits of conventional therapy are reduced; and or
* Critically ill patients at high risk of pulmonary embolism, not receiving medical thromboprophylaxis due to either increased risk of bleeding, active bleeding or heparin induced thrombocytopenia.

Since the Angel® Catheter is indicated for use in pregnant patients, patients who are pregnant may be included in this Registry after the proper risks and benefits have been assessed by the physician.

In summary, the Registry Event Schedule and data collection includes the following:

* Demographics and Current Medical Condition: Information collected to include demographics, medical condition and indication/s for use of the Angel® Catheter as recorded in the patient chart.
* Device Placement: Placement procedure data will be collected. If the catheter cannot be placed for some reason, no further follow up information will be collected on these patients.
* Angel® Catheter Indwelling experience: While the Angel® Catheter is in place during the patient's hospital stay, information regarding anticoagulation use (eCRF form #9), any complications, clinically significant PE, lower extremity DVT will be collected through three days after device retrieval, discharge from the hospital, or death, whichever occurs first.
* Device Retrieval: Information on ease of catheter retrieval and other key aspects will be collected.
* Registry Exit: Information about the patient's status at three days post device removal, death, or discharge from the hospital, whichever occurs first will be collected. The patient's date of discharge/transfer from the Critical Care Unit will also be collected.
* Anticoagulation Therapy: Information about the use of anticoagulation throughout the patient's observation period will be collected.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients in whom the Angel® Catheter is placed, or there has been an attempt to place.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry population will include all consecutive patients in whom the Angel® Catheter is placed, or there has been an attempt to place, at selected Registry sites.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Rate of averted PE | At the time of the pre-removal cavogram

SECONDARY OUTCOMES:
Incidence and seriousness of all device-related adverse events | While the Angel Catheter is in place, including the insertion and removal procedures (Up to 30 days)
Incidence and seriousness of deep vein thrombosis | From device placement through hospital discharge, death, or 3 days post-removal, whichever occurs first (Up to 33 days)
Incidence and seriousness of catheter-related thrombosis | From device placement through removal (Up to 30 days)
Incidence and seriousness of clinically significant PE | From device placement through hospital discharge, death, or 3 days post-removal, whichever occurs first (Up to 33 days)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Bunker, MD, Principal Investigator — Royal London Hospital
Locations (5):
- Germany (2):
  - Bremerhaven Reinkenheide Hospital, Bremersheide
  - University of Mannheim, Mannheim
- Ospendale Santa Maria di Loreto, Napoli, Italy
- United Kingdom (2):
  - Royal London Hospital, London
  - Royal Berkshire Hospital, Reading

IPD SHARING:
Plan to Share IPD: No